CLINICAL TRIAL: NCT01826266
Title: Phase I Evaluation of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Effects of a Double-Blind, Single Dose of PER977 Administered Alone, and Following a Single Dose of Edoxaban
Brief Title: Effects of a Double-Blind, Single Dose of PER977 Administered Alone, and Following a Single Dose of Edoxaban
Acronym: PER977-P1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Perosphere Pharmaceuticals Inc, a wholly owned subsidiary of AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: AMAG Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PER977-01-001; PER977-01-001 (Other: Perosphere)
Record Dates: First submitted 2013-04-03; First posted 2013-04-08 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2017-09

CONDITIONS: Anticoagulant Reversal; Reversal of Edoxaban Induced Anticoagulation
Keywords: PER977; Activated partial thromboplastin time; Assessment; D-dimer; Enrollment; Investigational drug; Investigational treatment; Period; Premature subject withdrawal; Prothrombin time; Randomization number; Study discontinuation; Study drug; Subject number; Study treatment; Thromboelastography-reaction time
MeSH Terms: interventions — PER977

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- PER977-Dose 1 (Placebo Comparator): Dose titration
  Interventions: Drug: PER977, Placebo
- PER977-Dose 2 (Placebo Comparator): Dose Titration
  Interventions: Drug: PER977, Placebo
- PER977-Dose 3 (Placebo Comparator): Dose Titration
  Interventions: Drug: PER977, Placebo
- PER977-Dose 4 (Placebo Comparator): Dose Titration
  Interventions: Drug: PER977, Placebo
- PER977-Dose 5 (Placebo Comparator): Dose Titration
  Interventions: Drug: PER977, Placebo
- PER977-Dose 6 (Placebo Comparator): Dose Titration
  Interventions: Drug: PER977, Placebo
- PER977-Dose 7 (Placebo Comparator): Dose Titration
  Interventions: Drug: PER977, Placebo

INTERVENTIONS:
Drug: PER977, Placebo
  Other Names: ciraparantag

SUMMARY:
PER977 monotherapy and co-administration following 60 mg edoxaban will have an acceptable safety and tolerability profile with no impact on pro-coagulant biomarkers. A dose of PER977 that reverses the effects of edoxaban on the pharmacodynamic (PD) biomarkers (point of care prothrombin time [PoC-PT]), and/or secondary biomarkers (thromboelastography reaction time [TEG-R]) will be identified.

DETAILED DESCRIPTION:
Normal subjects will be dosed with PER977 or placebo alone and 1 week later, they will be given a single dose of edoxaban followed in 3 hours by a single IV dose of PER977. The purpose is to show safety and tolerability of PER977 alone and when combined with a NOAC (edoxaban). The study will also provide some insight into the doses that may be required to reverse a steady state edoxaban.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18 to 45 years, inclusive
2. Laboratory values (chemistry, complete blood count coagulation assessments) and urinalysis performed during screening up to 21 days prior to administration of study treatment are within normal limits.
3. No clinically significant findings on 12-lead electrocardiogram (ECG) performed during screening.
4. Body mass index (BMI) 18 to ≤32 kg/m2, inclusive
5. Male subjects agree to use appropriate contraception (i.e., double barrier contraception such as a latex condom with spermicide with a female partner of child-bearing potential (a non-menopausal female who has not had one of the following: a) a hysterectomy (with or without oophorectomy), b) a bilateral oophorectomy without hysterectomy, or c) a medically documented ovarian failure) using a diaphragm or cervical cap or single barrier contraception if the female partner is using an intrauterine device or hormonal contraceptives or is sterilized; no barrier is required if the female partner has had a hysterectomy) when engaging in sexual activity during the course of the study. Moreover, male subjects should not donate sperm or attempt to impregnate a partner during the course of the study and for a period of 12 weeks following discharge from the study.
6. Female subjects of non-childbearing potential (a menopausal female with the above 3 definitions for menopause) agree to use two forms of non-hormonal contraceptive (e.g. barrier methods [condom or diaphragm]) or intrauterine device for the duration of the study and for 30 days following the completion of the study. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
7. Nonsmokers or nonusers of nicotine containing products within 3 months of dosing (occasional use of tobacco products within 30 days of dosing will be considered on a case-by-case basis)
8. Subjects must understand and agree to comply with the requirements of the study and they must be willing to sign the informed consent form indicating voluntary consent to participate in the study prior to initiation of screening or study related activities.

Exclusion Criteria:

1. History or current evidence of clinically significant cardiac, hepatic, renal, pulmonary, endocrine, neurologic, infectious, gastrointestinal, hematologic, or oncologic disease as determined by screening history, physical examination, laboratory test results or 12-lead ECG. History or current evidence of liver function tests greater than the upper limit of normal. History or current evidence of QTc Fridericia (QTcF) greater than normal (430±10 msec for males or 450±10 msec for females; average of three measurements).
2. History of unexplained syncope
3. Use of any drugs or substances known to be strong inhibitors or strong inducers of CYP3A4/5 transporters of p-glycoprotein within 28 days prior to the first dosing
4. History of major bleeding, trauma, surgical procedure of any type, or vaginal delivery within six months prior to screening
5. History of peptic ulcer, gastrointestinal bleeding (including hematemesis, melena, rectal bleeding) or bleeding from hemorrhoids within six months prior to screening
6. History of minor bleeding episodes such as epistaxis, rectal or hemorrhoidal bleeding (spots of blood on toilet paper) or gingival bleeding within 3 months prior to screening
7. Personal or family history of clotting disorder or abnormality, excessive bleeding, thrombovascular disease or any hematologic disorder involving platelets or clotting abnormalities or any condition requiring treatment with transfusions, anticoagulants or platelet inhibitors
8. Females with a history of dysfunctional uterine bleeding, including history of menorrhagia (heavy menstrual bleeding), metrorrhagia or polymenorrhea or current use of hormonal contraceptives.
9. Pregnant or breast-feeding
10. Male subjects with a history of hormone therapy within the 3 months prior to screening
11. Administration of any blood product or anticoagulant within 3 months prior to study entry or any non-steroidal anti-inflammatory drug or cyclooxygenase inhibitor within 2 weeks prior to screening
12. Taking any type of chronic medication within the 4 weeks prior to study entry
13. Positive serologic test for human immunodeficiency virus (HIV), Hepatitis C virus (HCV), or Hepatitis B surface antigen (HBsa)
14. Use of any of the following medications in the 4 weeks prior to study entry: rifampin, dronedarone, ketoconazole, verapamil, amiodarone, quinidine, clopidogrel, oral anticoagulants, or other agent known to interact with edoxaban
15. Donation of blood or blood products within 56 days prior to enrollment
16. Participation in any study with an investigational compound or device within 30 days prior to signing informed consent
17. Active drug, alcohol or nicotine use or dependence or any condition that, in the opinion of the Investigator, would interfere with adherence to study protocol

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety, tolerability, and plasma and urinary pharmacokinetics (PK) of a range of single intravenous (IV) doses of PER977 | 7 months

SECONDARY OUTCOMES:
Pharmacodynamic assessment | 2 days
  To determine the effect of escalating doses of PER977 on the reversal of edoxaban-induced anticoagulation

CONTACTS AND LOCATIONS:
Overall Officials: Robert Noveck, MD, PhD, Principal Investigator — Duke Clinical Research Unit
Locations (1):
- Duke Clinical Research, Unit 200, Durham, North Carolina, United States

REFERENCES:
- [Derived] Ansell JE, Bakhru SH, Laulicht BE, Steiner SS, Grosso MA, Brown K, Dishy V, Lanz HJ, Mercuri MF, Noveck RJ, Costin JC. Single-dose ciraparantag safely and completely reverses anticoagulant effects of edoxaban. Thromb Haemost. 2017 Jan 26;117(2):238-245. doi: 10.1160/TH16-03-0224. Epub 2016 Nov 17. PMID 27853809
- [Derived] Sciascia S, Lopez-Pedrera C, Cecchi I, Pecoraro C, Roccatello D, Cuadrado MJ. Non-vitamin K antagonist oral anticoagulants and antiphospholipid syndrome. Rheumatology (Oxford). 2016 Oct;55(10):1726-35. doi: 10.1093/rheumatology/kev445. Epub 2016 Feb 3. PMID 26843482
- [Derived] Ansell JE, Bakhru SH, Laulicht BE, Steiner SS, Grosso M, Brown K, Dishy V, Noveck RJ, Costin JC. Use of PER977 to reverse the anticoagulant effect of edoxaban. N Engl J Med. 2014 Nov 27;371(22):2141-2. doi: 10.1056/NEJMc1411800. Epub 2014 Nov 5. No abstract available. PMID 25371966